CLINICAL TRIAL: NCT00162045
Title: A Phase I-II, Open-Label, Multicenter Trial to Determine the Dosimetry and Safety of Technetium Tc99m Sestamibi in Pediatric Subjects
Brief Title: A Trial to Determine Radiation Exposure to Organs and Assess the Safety of CARDIOLITE® in Pediatric Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Qi Zhu, MD Senior Medical Director, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DuP 843-201
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Technetium Tc99m Sestamibi — Rest and/or stress SPECT imaging study

SUMMARY:
The purpose of this Phase I-II multicenter clinical trial is to establish dosimetry and safety profiles for CARDIOLITE® (Technetium Tc99m Sestamibi) in pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have been scheduled to undergo a clinically indicated rest or stress CARDIOLITE® MPI scan.
* Be able to comply with imaging requirements permitting completion of rest or stress CARDIOLITE® whole-body scans and SPECT imaging procedures without the use of sedation.

Exclusion Criteria:

* Have a terminal illness where expected survival is ≤6 months
* Have known clinically significant laboratory abnormalities (creatine, liver enzymes, platelet count).

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Determination of the absorbed radiation dose of Sestamibi in subjects will be evaluated at the end of the study through measurements of PK (blood and urine) up to 8 hours, dosimetry for 8 hours and image biodistribution for up to 8 hours | Following administration of Technetium Tc99m Sestamibi

SECONDARY OUTCOMES:
A determination of the safety of Sestamibi will be evaluated at the end of the study through adverse and serious adverse events reported and evaluating vital signs, ECGs, physical exams and laboratory tests for each subject | Following administration of Technetium Tc99m Sestamibi

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhu, MD, Study Director — Lantheus Medical Imaging
Locations (10):
- United States (7):
  - Jackson Memorial Hospital, Miami, Florida
  - Local Institution, Honolulu, Hawaii
  - University of Chicago Children's Hospital, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Wauwatosa, Wisconsin
- Local Institution, Vancouver, British Columbia, Canada
- Taiwan (2):
  - Local Institution, Changhua
  - Local Institution, Taichung

REFERENCES:
- [Derived] Azarbar S, Salardini A, Dahdah N, Lazewatsky J, Sparks R, Portman M, Crane PD, Lee ML, Zhu Q. A Phase I-II, Open-Label, Multicenter Trial to Determine the Dosimetry and Safety of 99mTc-Sestamibi in Pediatric Subjects. J Nucl Med. 2015 May;56(5):728-36. doi: 10.2967/jnumed.114.146795. Epub 2015 Apr 9. PMID 25858045